CLINICAL TRIAL: NCT06452511
Title: Comparing the Effect of Metformin vs. Pep2dia as an Adjunct to Letrozole on Ovulation Induction and Pregnancy Outcomes in Overweight Women With PCOS; A Randomized Controlled Open-Label Pilot Study
Brief Title: Comparing the Effect of Metformin vs. Pep2dia as an Adjunct to Letrozole on Ovulation Induction and Pregnancy Outcomes in Overweight Women With PCOS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Muhamed Ahmed Abdelmoaty Muhamed Alhagrasy (Other)
Responsible Party: Sponsor-Investigator, Muhamed Ahmed Abdelmoaty Muhamed Alhagrasy, lecturer and consultant at Obstetrics and Gynecology Department., Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Azhar524
Record Dates: First submitted 2024-06-01; First posted 2024-06-11 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: PCOS
Keywords: PCOS; Metformin; Pep2dia; overweight
MeSH Terms: conditions — Overweight | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Active Comparator): In the Metformin arm of this study, 50 overweight women with polycystic ovary syndrome (PCOS) who are experiencing infertility will participate. These participants will receive Letrozole for ovulation induction in combination with Metformin. The study will monitor these women to assess the efficacy of this treatment regimen on inducing ovulation and improving pregnancy outcomes. Participants will be closely observed for any side effects and their progress will be regularly evaluated to determine the effectiveness of Metformin as an adjunct therapy to Letrozole in this specific patient population.
  Interventions: Drug: Metformin
- Pep2Dia (Active Comparator): In the Pep2dia arm of this study, 50 overweight women with polycystic ovary syndrome (PCOS) who are experiencing infertility will participate. These participants will receive Letrozole for ovulation induction in combination with Pep2dia. The study will monitor these women to assess the efficacy of this treatment regimen on inducing ovulation and improving pregnancy outcomes. Participants will be closely observed for any side effects, and their progress will be regularly evaluated to determine the effectiveness of Pep2dia as an adjunct therapy to Letrozole in this specific patient population.
  Interventions: Drug: pep2dia

INTERVENTIONS:
Drug: Metformin — In the Metformin arm of this study, 50 overweight women with polycystic ovary syndrome (PCOS) and infertility will receive a combination treatment of Letrozole and Metformin. Letrozole, aimed at inducing ovulation, will be administered according to a specified dosage regimen, alongside Metformin, an insulin-sensitizing agent used to manage PCOS, prescribed at a specified dosage regimen. Participants will undergo regular monitoring to assess ovulation and pregnancy outcomes, involving baseline assessments of health status and fertility parameters, ongoing monitoring visits to track ovulation through ultrasound and hormone levels, and final evaluation of ovulation rates and pregnancy outcomes at the study's end. This arm seeks to determine the efficacy of Metformin as an adjunct to Letrozole in improving ovulation induction and pregnancy rates among overweight women with PCOS.
  Arms: Metformin
Drug: pep2dia — In the Pep2dia arm of this study, 50 overweight women diagnosed with polycystic ovary syndrome (PCOS) and experiencing infertility will receive a combination treatment of Letrozole and Pep2dia. Letrozole, utilized to induce ovulation, will be administered according to a specified dosage regimen, along with Pep2dia, a peptide-based therapy tailored to manage PCOS, prescribed at a specified dosage regimen. Participants will undergo regular monitoring to assess ovulation and pregnancy outcomes, involving baseline assessments of health status and fertility parameters, ongoing monitoring visits to track ovulation through ultrasound and hormone levels, and a final evaluation of ovulation rates and pregnancy outcomes at the conclusion of the study period. This arm seeks to ascertain the effectiveness of Pep2dia as an adjunct to Letrozole in enhancing ovulation induction and pregnancy rates among overweight women with PCOS.
  Arms: Pep2Dia

SUMMARY:
The goal of this clinical trial is to compare the effects of Metformin versus Pep2dia as adjunct treatments to Letrozole on ovulation induction and pregnancy outcomes in overweight women with polycystic ovary syndrome (PCOS). The main questions it aims to answer are:

Does Metformin improve ovulation rates more effectively than Pep2dia when used alongside Letrozole? Does Pep2dia enhance pregnancy outcomes compared to Metformin in this patient population?

Participants will:

Receive either Metformin or Pep2dia in addition to Letrozole. Undergo regular monitoring for ovulation and pregnancy outcomes. Researchers will compare the Metformin group to the Pep2dia group to see if there is a significant difference in ovulation and pregnancy rates between the two treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Anovulatory infertile women with PCOS for more than one year associated with overweight and seeking pregnancy.
2. Married women of reproductive age who lived with a husband and were sexually active.
3. Women with resistant to Letrozole.
4. Normal value of prolactin hormone.
5. Age group; 18-35 years
6. BMI ranging from 25 to 29 kg /m².
7. Standard parameters of the husband's semen
8. Diagnostic criteria for Rotterdam diagnosis of polycystic ovary syndrome:

Two of the following three criteria are required:

* Oligoovulation or Anovulation
* Hyperandrogenism: Clinical (hirsutism or less commonly male pattern alopecia) or Biochemical (raised free androgen index (FAI) or free testosterone).
* Polycystic ovaries on ultrasound (Christ et al., 2023).

Exclusion Criteria:

1. Hypersensitivity to letrozole, metformin or pep2dia.
2. Obese women with BMI ≥29 kg/m² or women with BMI <25 kg/m².
3. FSH above 11 mg.
4. Any other cause of infertility other than anovulation due to overweight as uterine factor, tubal factor, male factor, ovarian pathology or endometriosis.
5. Any medical disorder that may affect pregnancy or systemic disease (cardiovascular, renal, hepatic, CNS diseases and hypo or hyperthyroidism)
6. Missed patient
7. Discontinuation of drug due to its side effects

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study will include only female participants. The eligibility criteria specify that all participants must be women diagnosed with polycystic ovary syndrome (PCOS) who are experiencing infertility. These women should be overweight, as defined by a body mass index (BMI) within the specified range for the study. No male participants will be included in this trial.
Enrollment: 100 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate: | 6 months
  detected by positive pregnancy test in serum (Chemical pregnancy) or presence of intrauterine gestational sac (Clinical pregnancy)

SECONDARY OUTCOMES:
Ovulation rate: | 6 months
  detected by folliculometry and midluteal progesterone in serum (higher than 3 ng/mL)
Menstrual cycle regulation | 6 months
  Detection of regulation of the menstrual cycle that is not regular in patients with PCOS assessed as cycle length 21-35 days.
Side effects of both agents | Throughout the study time (up to 1 year).
  Monitoring and recording of any adverse effects experienced by participants during the study period
Ongoing pregnancy rate after the first trimester | first 13 weeks in pregnancy.
  Assessment of the proportion of pregnancies that progress beyond the first trimester

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Hussein University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
In accordance with the decision not to share individual participant data (IPD), strict measures will ensure confidentiality. Data collection will maintain anonymity, with unique identifiers replacing personal details. All data, from demographics to outcomes, will be securely stored in encrypted databases accessible only to authorized personnel. Individual participant data won't be shared externally; aggregate data may be shared while protecting privacy. Participants will be fully informed, addressing any concerns on data privacy during consent and throughout. The study protocol will undergo ethical review, ensuring compliance with confidentiality standards. Regular audits will monitor compliance with data security, promptly addressing breaches. These measures uphold participant confidentiality while investigating Metformin and Pep2dia effects on overweight women with PCOS undergoing Letrozole-induced ovulation.